CLINICAL TRIAL: NCT06412289
Title: A Prospective, Randomized, Multicentric and Single-blinded Study on Accuracy and Safety of Ultrasound (US) Guided Percutaneous Needle Biopsy of Peripheral Lung Lesion Compared With Computed TomogrAphy (CT) Guided Needle Biopsy
Brief Title: Comparison of the Diagnostic Accuracy: US-guided Percutaneous Lung Biopsies vs CT-guided in Peripheral Lung Lesions
Acronym: SULTAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Mario Tamburrini, Principal investigator, University Hospital of Ferrara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 648/2023/Sper/AOUFe
Record Dates: First submitted 2024-04-29; First posted 2024-05-14 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Peripheral Lung Lesions

STUDY DESIGN:
Who Masked: Investigator
Masking Description: anatomopathologist is blinded about the procedure which has been executed
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- US-guided percutaneous needle biopsy (Experimental): Patients who are randomized into this arm will undergo US-percutaneous needle biopsy to sample the lesion. A convex probe is used to visualize the lung lesion and execute the percutaneous procedure. One hour after the end of the procedure, a chest x-ray is requested.
  Interventions: Diagnostic Test: US-GUIDED PERCUTANEOUS LUNG NEEDLE BIOPSY
- CT-guided percutaneous needle biopsy (Experimental): Patients who are randomized into this arm will undergo CT-percutaneous needle biopsy. The procedure is done by using a CT scan to measure and identify the right point where the percutaneous biopsy will be executed. One hour after the end of the procedure, a chest x-ray is requested.
  Interventions: Diagnostic Test: CT-GUIDED PERCUTANEOUS LUNG NEEDLE BIOPSY

INTERVENTIONS:
Diagnostic Test: US-GUIDED PERCUTANEOUS LUNG NEEDLE BIOPSY — The ultrasound investigation will be conducted using the ultrasound machine supplied to the Center involved in the trial and usually used in eTTNA procedures. Before the procedure, the vital signs of the patient will be noted and each operator will choose the most appropriate position for the sampling, based on the location of the lesion. The thoracic area to biopsy will then be defined and then there will be the setting of the sterile field. At this point, local anesthesia with a maximum of 20ml of 2% lidocaine will be administrated, marking down this time as the time of the beginning of the procedure. 18 Gauge needles will be used to collect the sample. For each patient, there will be collected a minimum number of one and a maximum number of three bioptic sampling .
  Arms: US-guided percutaneous needle biopsy
Diagnostic Test: CT-GUIDED PERCUTANEOUS LUNG NEEDLE BIOPSY — The CT scan will be performed using the CT machinery equipped by the Center involved in the trial and usually used for the tTTNA procedures. Before the procedure, the vital signs of the patient will be noted and each operator will choose the most appropriate position for the sampling, based on the location of the lesion. The thoracic area to biopsy will then be defined and then there will be the setting of the sterile field. At this point, local anesthesia with a maximum of 20ml of 2% lidocaine will be administrated, marking down this time as the time of the beginning of the procedure. 18 Gauge needles will be used to collect the sample. For each patient, there will be collected a minimum number of one and a maximum number of three bioptic sampling .
  Arms: CT-guided percutaneous needle biopsy

SUMMARY:
A non-sponsored prospective randomized single-blind national multicenter interventional study which aims to compare the diagnostic accuracy between US-guided percutaneous lung needle biopsies and CT-guided in peripheral lung lesions. Secondary endpoints are:

* onset of number and type of complications during and after the procedure, within the first three hour;
* exposition to ionizing radiation, in milligray(mGy);
* patient comfort during the procedure;
* duration of the procedure,

DETAILED DESCRIPTION:
Peripherical pulmonary lesions without endobronchial lesions (LPP) are nowadays more and more frequently found in clinical practice, and it's only assumable that this tendency will keep growing in the future, alongside the increasing use of thoracic CT scanning and the proven efficacy in lung cancer screening. Even though most of these lesions are benign, it's still important to be able to identify neoplastic lesions in an early stage.

The gold standard for diagnosis definition is biopsy, which can be performed by four paths: surgery, transbronchial endoscopy (TBB), endobronchial endoscopy (EBB) or percutaneous (TTNA).

Surgical option is the most reliable one in terms of diagnostic yield, at the expense of an increased risk of complications, post-operative recovery in hospital staying and costs, compared with the other three procedures; due to the safety and diagnostic yield of TBB, EBB and TTNA, the surgical approach, just for the purpose of diagnosis, resulted in a secondary choice in the diagnostic flowchart of LPP. In addiction, given the high probability of the benign nature of the LPP, the choice of a less invasive approach in the diagnostic phase is even more reasonable. Even though technology really improved the diagnostic yield of LPP, overall sensibility is around 70-80%, influenced by many factors such as: localization and extension of the lesion, presence of bronchus sign, sampling techniques and procedural errors. The incidence of complications for this type of sampling, mostly presented by pneumothorax, is around 4%.

The TTNA is a largely used procedure for diagnosing LPP and it can be conducted using both a CT guided and an ultrasound guided approach, as long as the lesion is located in direct contact with the thoracic wall. CT scan guide has the perk of giving a more precise view of: densitometric feature of the lesions, their location and the connections with the anatomical structures surrounding them. LPP CT guided TTNA (tTTNA) can reach a diagnostic yield of 98% in case of an experienced operator, where ultrasound guided reaches about 93.4%, only slightly inferior to the prior one. Both tTTNA and ultrasound guided percutaneous transthoracic biopsy (eTTNA) are useful techniques not only for pulmonary parenchymal diseases but also in case of pleural lesions, allowing simultaneous sampling and visualization of the lesions in exam.

Peripheric pleural lesions can also be approached via thoracoscopy (both medical and surgical) with a diagnostic efficiency between 91-95% for malignant lesions and 100% for Tuberculosis-related lesions. However, the high risk of complications after the procedure, the duration of hospitalization post-surgery and the costs, suggest choosing between eTTNA and tTTNA as the very first diagnostic step in pleural lesions as well. Moreover, the diagnostic yield of tTTNA and eTTNA is respectively of 89% and 90%.

Both eTTNA and tTTNA demonstrated a good ability in distinguishing between benign and malignant lesions. In the latter case, collecting a representative enough sample allows the appropriate immunohistochemical phenotyping and genetic sequencing of it, enabling to make targeted therapeutical choices according to the current Guidelines.

Literature suggests that the number of bioptic steps necessary to obtain an adequate diagnostic sample is of three steps, where an upper number of them would increase the risk of complications despite an almost equal diagnostic efficiency. Principal complications of percutaneous sampling, common to both the approaches, are pneumothorax and minor bleeding (not requiring blood transfusion) In literature there are no clear indications about which of these two methods is better in case of lesions touching the pleural surface, therefore approachable with both tTTNA and eTTNA; in everyday clinical practice the choice is mostly driven by the availability of each technique in the Center of expertise. Also, from the literature that could be gathered, there is no prospective comparison between ultrasound-guided and CT-guided needle biopsy of peripheric pulmonary lesion touching the thoracic wall.

Nonetheless, a trial retrospectively analyzed both ultrasound-guided and CT-guided sampling of thoracic lesions touching the wall and it enlightened that the complications rate was minor for the ultrasound-guided approach: respectively 3.3% and 24%. Even more, differently from the tTTNA, eTTNA doesn't expose the patients to any ionizing radiation and it allows to avoid artefacts deriving from respiratory movements and the ribs' interposition.

On this ground of observations, we present the following trial, which would be the first prospective one to compare the diagnostic accuracy between the two approaches (tTTNA and eTTNA) for diagnosing peripheric pulmonary lesions touching the thoracic wall.

The trial's goal is comparing the diagnostic yield of ultrasound-guided vs CT-guided histological sampling of peripheric pulmonary lesions touching the thoracic wall.

All patients must, therefore, have carried out recent blood tests (within one month before the procedure) routine including: complete blood count, international normalized ratio(INR), activated partial thromboplastin time(aPTT), prothrombin time(PT).

When taking charge of the patient, the inclusion and exclusion criteria will be verified. The patient candidate for the procedure signs the informed consent to the study in the presence of the local coordinator or co-investigator. The coordinator or co-investigator will proceed with the randomization (through random numbers generated by a computer) to perform ultrasound-guided or CT-guided sampling, which will be scheduled with the usual technical times of each individual participating Center.

Each patient will be assigned a progressive number/code for anonymization purposes to be used in the electronic Case Report Form(eCRF). The diagnostic procedures will be carried out in the Respiratory Endoscopy and Radiology rooms where TTNAs are usually carried out. The ultrasound investigation will be conducted using the ultrasound machine supplied to the Center involved in the trial and usually used in eTTNA procedures.

The CT scan will be performed using the CT machinery equipped by the Center involved in the trial and usually used for the tTTNA procedures.

Before the procedure, the vital signs of the patient will be noted and each operator will choose the most appropriate position for the sampling, based on the location of the lesion. The thoracic area to biopsy will then be defined and then there will be the setting of the sterile field. In accordance to the guide-lines the patient should not be sedated if possible. At this point, local anesthesia with a maximum of 20ml of 2% lidocaine will be administrated, marking down this time as the time of the beginning of the procedure.

18 Gauge needles will be used to collect the samples, since this size allows a good balancing between risk of complication and diagnostic yield. For each patient, there will be collected a minimum number of one and a maximum number of three bioptic sampling. The sample will be stored and preserved inside specific containers to allow optimal transfer to the Pathology laboratories, based on the directions of the laboratory itself and the usual procedure of the involved Center.

Once the procedure is done, the patient will remain in the involved Center for a period of observation of at least three hours. During this time, the patient will be monitored through vital signs and the occurrence of any complication. After one hour from the procedure, a thoracic X-Ray examination will be taken, preferably in orthostatism, in both inhale and exhale. The management of any possible complication will be carried out as part the singular Center's practice, in agreement with the latest Guide Lines regarding the matter.

In the case of the impossibility of the technical use of the procedure assign to the singular patient by the randomization, the patient will be excluded from the trial and will carry on the diagnostic iter according to the usual clinical practices.

The onset of complications will be registered during the patients' monitoring process, which will last for the three hours following the procedure. All the participant patients will be informed about the possible late-onset complications after the procedure and about the necessity of coming back to the hospital in case of the occurrence of any symptoms, such as dyspnea, chest pain, hemoptysis/bloody sputum.

The anatomopathologist will receive the samples without the indication of the methodic used for the biopsy. The pathologist will, then, pronounce judgment un: 1) adequacy of the samples for the purpose of the diagnosis 2) where indicated, the suitability for a full histological molecular analysis. Once the diagnosis is given, the local coordinator or the co-investigators will communicate the result to the patient as soon as possible, in order to address the patient to the currently most appropriated diagnostic-therapeutic pathway.

The tissue sample will be submitted to the pathologist along with a form containing personal data, anamnesis, clinical suspicion, the sample topography and the trial code. In order to preserve the double-blind criteria in the anatomopathological reporting, all the requests coming from a center will submitted after the name of the local coordinator. The pathologist will report the resulting diagnosis to his center's the coordinator via email and only then it will be possible to move forward to the unblinding. Enrolled patients will be entered in an eCRF file, shared exclusively between the interventional operators. Therefore, the patients will be addressed to the best diagnostic-therapeutic program available at the time, according to the most recent guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Willingness and ability to provide free and informed consent. Age older then 18 years old.
* Peripheric pulmonary lesions adherent to the thoracic wall in CT scans with indication to typing

Exclusion Criteria:

* Inability to provide free and informed consent, in the absence of an available legal guardian.
* Age younger then 18 years old.
* Terminal neoplastic diseases/ palliative care patients.
* Patients with one lung, anatomical of functional.
* Severe non-treatable blood clothing disfunctions.
* Severe organ failure (pulmonary, renal, hepatic or cardiac).
* Women in state of pregnancy.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2024-03-08 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Rate of diagnostic samples vs rate of non diagnostic samples assessed by the histological reports, detecting the ones positive for malignant neoplasm or specific benign process out of the totality of procedures for both US-guided and CT-guided biopsy | 1 month
  For diagnostic sampling is meant the ability to diagnose a malignant neoplasm or a specific benign process (such as benignant neoplasia, granulomatous inflammation). For nondiagnostic sample is meant the finding of a non-specific benign process or that the sample is not adequate/sufficient. For benign non-specific is meant a histological diagnosis suggesting a benign process without any evidence of malignancy but that does not give the specific information to achieve a definitive diagnosis. In any case that does not include a diagnostic confirmation of a non-specific benign lesion by a surgical approach, TTNA will be considered a true negative only after a follow-up documenting a downsizing of at least 20% in the major axial diameter or a stability in sizing for at least one year from the lesion itself.

SECONDARY OUTCOMES:
Rate of complications that can be occur during the procedures assessed by physiological parameter, VAS scale, radiography | 3 hours
  The data about number and the type of complications during and after the procedure will be collected to calculate the rate of complications for both US-guided and CT-guided biopsies. The investigator will evaluate the pain by VAS scale which goes from 0 (no pain) to 10 (worst pain possible). The physiological parameters will be checked during the procedure and within three hours after the procedure. The patient will undergo radiography to check one hour after the procedure.
Amount of Ionizing radiation to which the patient is exposed calculated in mGy | 1 hour
  During each procedure of CT-guided biopsy the investigators will obtain information about the amount of ionizing radiation to which the patient is exposed and this will be reported in mGy.
Comfort of the patient during the procedure assessed by Visual Analog Pain Scale(VAS scale) | 1 hour
  The patient will be asked about the discomfort related to the procedure by VAS scale, which goes from 0 (extreme discomfort-absence of comfort) to 100 (extreme comfort-absence of discomfort)
Duration of the procedure in seconds | 1 hour
  The duration of each procedure (from the time of the local anesthesia for the time of the extraction of the last biopsy)will be calculated and reported in seconds
Rate of sample suitable for next-generation sequencing(NGS) analysis based on percentage of neoplastic cell in samples | 1 month
  Regarding malignant lesions, for those eligible to molecular target therapy, samples will be divided based on the percentage of neoplastic cells in the sample (T%) in T% >20% (suitable for NGS analysis) and T% <20% (non-suitable for NGS analysis)

CONTACTS AND LOCATIONS:
Overall Officials: Mario Tamburrini, Dr., Principal Investigator — Arcispedale Sant'Anna
Locations (2):
- Italy (2):
  - UO Pneumologia AOSP-AUSL, Ferrara
  - UOC Pneumologia - Azienda ospedaliera A. Cardarelli, Napoli

REFERENCES:
- [Background] Asano F. Advanced bronchoscopy for the diagnosis of peripheral pulmonary lesions. Respir Investig. 2016 Jul;54(4):224-9. doi: 10.1016/j.resinv.2015.11.008. Epub 2016 Mar 2. PMID 27424820
- [Background] Wang B, Zhong F, An W, Liao M. The diagnostic value of CT-guided percutaneous puncture biopsy of pulmonary ground-glass nodules: a meta-analysis. Acta Radiol. 2023 Apr;64(4):1431-1438. doi: 10.1177/02841851221137693. Epub 2022 Nov 15. PMID 36380521
- [Background] Baratella E, Cernic S, Minelli P, Furlan G, Crimi F, Rocco S, Ruaro B, Cova MA. Accuracy of CT-Guided Core-Needle Biopsy in Diagnosis of Thoracic Lesions Suspicious for Primitive Malignancy of the Lung: A Five-Year Retrospective Analysis. Tomography. 2022 Nov 25;8(6):2828-2838. doi: 10.3390/tomography8060236. PMID 36548528
- [Background] Criner GJ, Eberhardt R, Fernandez-Bussy S, Gompelmann D, Maldonado F, Patel N, Shah PL, Slebos DJ, Valipour A, Wahidi MM, Weir M, Herth FJ. Interventional Bronchoscopy. Am J Respir Crit Care Med. 2020 Jul 1;202(1):29-50. doi: 10.1164/rccm.201907-1292SO. PMID 32023078
- [Background] Yamamoto N, Watanabe T, Yamada K, Nakai T, Suzumura T, Sakagami K, Yoshimoto N, Sato K, Tanaka H, Mitsuoka S, Asai K, Kimura T, Kanazawa H, Hirata K, Kawaguchi T. Efficacy and safety of ultrasound (US) guided percutaneous needle biopsy for peripheral lung or pleural lesion: comparison with computed tomography (CT) guided needle biopsy. J Thorac Dis. 2019 Mar;11(3):936-943. doi: 10.21037/jtd.2019.01.88. PMID 31019783
- [Background] Ikezoe J, Sone S, Higashihara T, Morimoto S, Arisawa J, Kuriyama K. Sonographically guided needle biopsy for diagnosis of thoracic lesions. AJR Am J Roentgenol. 1984 Aug;143(2):229-34. doi: 10.2214/ajr.143.2.229. PMID 6611048
- [Background] Niu XK, Bhetuwal A, Yang HF. CT-guided core needle biopsy of pleural lesions: evaluating diagnostic yield and associated complications. Korean J Radiol. 2015 Jan-Feb;16(1):206-12. doi: 10.3348/kjr.2015.16.1.206. Epub 2015 Jan 9. PMID 25598692
- [Background] Koegelenberg CF, Irusen EM, von Groote-Bidlingmaier F, Bruwer JW, Batubara EM, Diacon AH. The utility of ultrasound-guided thoracentesis and pleural biopsy in undiagnosed pleural exudates. Thorax. 2015 Oct;70(10):995-7. doi: 10.1136/thoraxjnl-2014-206567. Epub 2015 May 21. PMID 25997433
- [Background] Knox D, Halligan K. Case series of trans-thoracic nodule aspirate performed by interventional pulmonologists. Respir Med Case Rep. 2021 Feb 2;32:101362. doi: 10.1016/j.rmcr.2021.101362. eCollection 2021. PMID 33665077
- [Background] Lim C, Lee KY, Kim YK, Ko JM, Han DH. CT-guided core biopsy of malignant lung lesions: how many needle passes are needed? J Med Imaging Radiat Oncol. 2013 Dec;57(6):652-6. doi: 10.1111/1754-9485.12054. Epub 2013 Apr 1. PMID 24283552
- [Background] Manhire A, Charig M, Clelland C, Gleeson F, Miller R, Moss H, Pointon K, Richardson C, Sawicka E; BTS. Guidelines for radiologically guided lung biopsy. Thorax. 2003 Nov;58(11):920-36. doi: 10.1136/thorax.58.11.920. No abstract available. PMID 14586042
- [Background] Moore W, Sawas A,Lee C,Ferretti J,
- [Background] Kim D, Han JY, Baek JW, Lee HY, Cho HJ, Heo YJ, Shin GW. Effect of the respiratory motion of pulmonary nodules on CT-guided percutaneous transthoracic needle biopsy. Acta Radiol. 2023 Jul;64(7):2245-2252. doi: 10.1177/02841851221144616. Epub 2022 Dec 27. PMID 36575592
- [Background] DiBardino DM, Yarmus LB, Semaan RW. Transthoracic needle biopsy of the lung. J Thorac Dis. 2015 Dec;7(Suppl 4):S304-16. doi: 10.3978/j.issn.2072-1439.2015.12.16. PMID 26807279